CLINICAL TRIAL: NCT00882063
Title: An Open Label, Multicenter Phase I/II Study To Evaluate Safety and Efficacy of P276-00 in Subjects With Relapsed and/or Relapsed/Refractory Multiple Myeloma
Brief Title: Study To Evaluate Safety and Efficacy of P276-00 in Subjects With Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/15/07
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P276-00 (Experimental): Starting dose level of P276-00 is 50 mg/m2/day. The drug will be administered intravenously in 200 ml of 5% dextrose (D5W) over a period of 30 min. Subjects will be enrolled at different dose levels of P276-00 to determine maximum tolerated dose of P276-00.
  Interventions: Drug: P276-00

INTERVENTIONS:
Drug: P276-00 — Subjects will be enrolled at different dose levels of P276-00 to determine maximum tolerated dose of P276-00.Starting dose level of P276-00 is 50 mg/m2/day to be administered intravenously in 200 ml of 5% dextrose (D5W) over a period of 30 min from day 1 to day 5 every 21 days. This constitutes one cycle of P276-00. Six such cycles will be administered to subjects.

SUMMARY:
The purpose of this study is to determine safety of P276-00 in patients with advanced multiple myeloma and whether P276-00 is effective in the treatment of advanced cases of multiple myeloma.

DETAILED DESCRIPTION:
This is an open label multicenter study of P276-00 in subjects with Relapsed and/or Relapsed/Refractory Multiple Myeloma. Cohort of 3 subjects will be enrolled at starting dose of P276-00 which is 50 mg/m2/day to be given intravenously from day 1 to day 5 every 21 days. This 21 day administration constitutes one cycle of P276-00. Six such cycles will be administered to the subjects. If the dose is well tolerated then next cohort will be enrolled at higher dose level of P276-00 till maximum tolerated dose is determined. Safety assessment will be repeated at regular interval and efficacy assessment will be repeated during every cycles.After the subject completes 6 cycles, there will be a follow-up visit after 4 weeks (+1 week) of study completion.Subjects who have stable disease or who have responded (MR, PR or CR) after completion of the 6 cycles will be given the option to continue treatment for a maximum of 12 cycles or until they are deemed to have progressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects previously diagnosed with multiple myeloma based either on the standard diagnostic criteria or the International Myeloma Foundation (IMF) diagnostic criteria as defined in Appendix A.
2. Subjects must have relapsed and/or relapsed/refractory disease after at least 2 prior lines of therapy as defined in Appendix D.
3. Monoclonal protein in the serum of > or = 1 g/dL or monoclonal light chain in the urine protein electrophoresis of > or = 200 mg/ 24 hours, or measurable light chains by free light chain assay of > or = 10 mg/dL, or measurable plasmacytoma.
4. Age > or = 18 years at the time of signing the informed consent form
5. ECOG performance status < or = 2
6. Life expectancy > or = 3 months
7. Subjects must have the following laboratory parameters:

   * Hemoglobin > or = 8.0 gm/dL
   * Absolute Neutrophil Count (ANC) > or = 1000 cells/mm3
   * Platelets count > or = 50,000/mm3
   * Serum SGOT/AST <3.0 x institutional upper limits of normal (ULN)
   * Serum SGPT/ALT <3.0 x institutional upper limits of normal (ULN)
   * Serum creatinine <2.5mg/dL
   * Serum total bilirubin <1.5 x institutional upper limits of normal (ULN)
8. Woman of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months) with a negative serum pregnancy test. In addition, all sexually active women of childbearing potential and men agreeing to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilised.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Subjects having received radiotherapy, immunotherapy, chemotherapy and/or biological agents like G-CSF in the 4 weeks prior to day 1 of study drug administration or have not recovered (grade < or = 1) from adverse effects of such therapy received prior to 4 weeks
2. Subjects having received any other investigational agents within 4 weeks prior to the date of enrolment or have not recovered from adverse effects of the investigational agent received prior to 4 weeks.
3. History of allergic reactions attributed to compounds of similar chemical composition to P276-00.
4. Subjects with a history of myocardial infarction or uncontrolled cardiac dysfunction during the previous 6 months.
5. Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer or any other cancer for which the subject has been disease-free for at least 3 years.
6. Subjects with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, cardiac ejection fraction < 40%, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
7. Women who are pregnant or nursing
8. Subjects known to be seropositive for the human immunodeficiency virus or any history or evidence from physical examination of HIV infection.
9. Subjects requiring the use of concomitant medications that prolong the QT/QTc interval and/or are known to cause Torsades de Pointes (TdP).
10. Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of P276-00 in subjects with relapsed and/or relapsed/refractory Multiple Myeloma | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu Parikh, M.D., Study Director — Vice President- Clinical Research (R & D), Nicholas Piramal Research Centre
Locations (5):
- India (5):
  - Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - Shatabdi Superspeciality Hospital, Nashik, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, Delhi, National Capital Territory of Delhi
  - Institute Rotary Cancer Hospital,All India Institute Of Medical Sciences(AIIMS), New Delhi, New Delhi
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata, West Bengal